CLINICAL TRIAL: NCT05075668
Title: Continuous Positive Airway Pressure Therapy Via Conventional CPAP Face Mask Versus High Flow Nasal Cannula in OSA Patients on the First Postoperative Night- a Pilot Randomised Study
Brief Title: Efficacy of HFNC as an Alternative to CPAP Therapy in Surgical Patients With Suspected Moderate to Severe OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Tsai Fung Chen, Consultant, Department of Anaesthesia & Surgical Intensive Care, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2142
Record Dates: First submitted 2019-11-13; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: OSA
Keywords: CPAP therapy; High flow nasal cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- OSA support via CPAP face mask (Active Comparator): Auto-titrated according to the settings made by sleep physicians, FiO2 0.21
  Interventions: Device: CPAP face mask
- OSA support via HFNC at 20 L/min (Active Comparator): High flow nasal insufflation of air (FiO2 0.21) at 20 L/min
  Interventions: Device: High flow nasal cannula (HFNC)
- OSA support via HFNC at 30 L/min (Active Comparator): High flow nasal insufflation of air (FiO2 0.21) at 30 L/min
  Interventions: Device: High flow nasal cannula (HFNC)
- OSA support via HFNC at 40 L/min (Active Comparator): High flow nasal insufflation of air (FiO2 0.21) at 40 L/min
  Interventions: Device: High flow nasal cannula (HFNC)

INTERVENTIONS:
Device: CPAP face mask — Two types of CPAP therapy for OSA support are compared; CPAP face mask vs HFNC at different flow rates
  Arms: OSA support via CPAP face mask
Device: High flow nasal cannula (HFNC) — Two types of CPAP therapy for OSA support are compared; CPAP face mask vs HFNC at different flow rates
  Other Names: Optiflow™ High Flow therapy; Fisher and Paykel
  Arms: OSA support via HFNC at 20 L/min; OSA support via HFNC at 30 L/min; OSA support via HFNC at 40 L/min

SUMMARY:
High flow, humidified, temperature-regulated nasal insufflation is not a new concept. It is used widely in the treatment of hypoxaemic respiratory failure in critically ill patients, as an alternative to non-invasive positive ventilation via face or nasal mask. Recently, its use has been extended to the perioperative setting for pre-oxygenation and prolonging apnoeic time to desaturation. Both CPAP and high flow nasal cannula insufflation devices are licensed for use clinically in Singapore. We conduct this pilot study because its perioperative use in our adult OSA population is currently not well-defined.

DETAILED DESCRIPTION:
Continuous positive airway pressure (CPAP) therapy is the only treatment for obstructive sleep apnoea (OSA) shown to reduce its long-term adverse effects on the cardiovascular system. However, due to difficult patient-mask interface and discomfort, compliance rate amongst patients with OSA is low, and reported to be only between 20-50%. High flow, humidified, temperature-regulated nasal cannula insufflation (of air or oxygen) is a well-documented and safe treatment in intensive care, paediatrics and respiratory medicine for patients with hypoxaemic respiratory failure. Its use in adult patients with obstructive sleep apnoea, especially in the perioperative setting is not well studied. Our hospital has a ''fast-track'' protocol for OSA patients who require surgery. They are started on CPAP therapy 2 to 5 days prior to surgery and in the immediate post operative period (ie. perioperatively). If these patients are non-compliant to the CPAP mask device, high flow nasal insufflation is a possible alternative treatment. We aim to randomise these patients into 4 groups, receiving conventional CPAP face mask or high flow nasal cannula at 3 flow rates, and study them with respect to incidence and number of documented desaturations. In addition, patient satisfaction, compliance to device and any adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-85 years old presenting for elective surgery.
* Suspected/possible OSA patients who are enrolled in the "fast-track OSA protocol" in the pre-assessment clinic
* Patients started on CPAP therapy at least one day pre-operatively
* Patients who are admitted to the High Dependency unit for postoperative monitoring.

Exclusion Criteria:

* Patients with nasal obstruction.
* Patients undergoing nasal or facial surgery, or surgery to treat OSA (eg. uvulopalatopharyngoplasty).
* Patients who already require a higher oxygen concentration (FiO2 > 0.21) preoperatively.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with documented desaturations (defined as >4% drop from baseline) | 10 hours (between 10pm on first postoperative night and 8am the following day)
  Number of documented desaturations (defined as >4% below baseline) in OSA patients who receive CPAP face mask or high flow nasal insufflation on the first postoperative night

SECONDARY OUTCOMES:
Number of participants who need for supplemental oxygen and/ or the need for other interventions to reverse the desaturations. | 10 hours (between 10pm on first postoperative night and 8am the following day)
  Need for supplemental oxygen and/or the need for other interventions to reverse desaturations in OSA patients who receive CPAP face mask or high flow nasal insufflation on the first postoperative night
Patients' perceptions of the comfort of each device on scale of 0 to 100 | 10 hours (between 10pm on first postoperative night and 8am the following day)
  The patients' perceptions of the comfort of CPAP face mask and/ or high flow nasal insufflation
Number of participants with any adverse effects of the applied therapy in the immediate postoperative setting. | 10 hours (between 10pm on first postoperative night and 8am the following day)
  OSA patients who receive CPAP face mask or high flow nasal insufflation on the first

CONTACTS AND LOCATIONS:
Overall Officials: Fung Chen Tsai, MMED (Anaes), Principal Investigator — Changi General Hospital, SingHealth
Locations (1):
- Changi General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Gotera C, Diaz Lobato S, Pinto T, Winck JC. Clinical evidence on high flow oxygen therapy and active humidification in adults. Rev Port Pneumol. 2013 Sep-Oct;19(5):217-27. doi: 10.1016/j.rppneu.2013.03.005. Epub 2013 Jul 8. PMID 23845744
- [Background] Zhang J, Lin L, Pan K, Zhou J, Huang X. High-flow nasal cannula therapy for adult patients. J Int Med Res. 2016 Dec;44(6):1200-1211. doi: 10.1177/0300060516664621. Epub 2016 Oct 3. PMID 27698207
- [Background] McGinley BM, Patil SP, Kirkness JP, Smith PL, Schwartz AR, Schneider H. A nasal cannula can be used to treat obstructive sleep apnea. Am J Respir Crit Care Med. 2007 Jul 15;176(2):194-200. doi: 10.1164/rccm.200609-1336OC. Epub 2007 Mar 15. PMID 17363769
- [Background] Nilius G, Wessendorf T, Maurer J, Stoohs R, Patil SP, Schubert N, Schneider H. Predictors for treating obstructive sleep apnea with an open nasal cannula system (transnasal insufflation). Chest. 2010 Mar;137(3):521-8. doi: 10.1378/chest.09-0357. Epub 2009 Dec 1. PMID 19952061
- [Background] Sowho MO, Woods MJ, Biselli P, McGinley BM, Buenaver LF, Kirkness JP. Nasal insufflation treatment adherence in obstructive sleep apnea. Sleep Breath. 2015 Mar;19(1):351-7. doi: 10.1007/s11325-014-1027-4. PMID 25015548
- [Background] Nilius G, Franke KJ, Domanski U, Schroeder M, Ruhle KH. Effect of APAP and heated humidification with a heated breathing tube on adherence, quality of life, and nasopharyngeal complaints. Sleep Breath. 2016 Mar;20(1):43-9. doi: 10.1007/s11325-015-1182-2. Epub 2015 May 10. PMID 25957615